CLINICAL TRIAL: NCT01754870
Title: HO11415: Phase II Study of Bendamustine and Rituximab Induction Chemoimmunotherapy Followed by Maintenance Rituximab (Rituxan®) and Lenalidomide (Revlimid®) in Relapsed and Refractory Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
Brief Title: Phase II Study of Bendamustine and Rituximab Induction Chemoimmunotherapy Followed by Maintenance Rituximab (Rituxan®) and Lenalidomide (Revlimid®) in Relapsed and Refractory Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO11415; 2012-0639 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); NCI-2013-00905 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2012-11-27; First posted 2012-12-21 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2015-07

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine + Rituximab-->Rituximab and Lenalidomide (Experimental): Induction chemoimmunotherapy:
  * Bendamustine 70 mg/m2 IV days 1 & 2 every 28 days X 6 cycles
  * Rituximab 500 mg/m2 IV day 1 every 28 days X 6 cycles (375 mg/m2 IV cycle 1 only, day 1 or 2)
  Maintenance phase:
  * Rituximab 375 mg/m2 IV on day 1 of every odd-numbered 28 day cycle for a maximum of 12 doses during the maintenance phase.
  * Lenalidomide 5 mg orally daily on days 1-28 of each 28-day cycle for 24 cycles (maintenance cycles 1-24); dose escalation to 10 mg orally daily will be allowed at the start of cycle 2 or at the start of any subsequent cycle in subjects with acceptable toxicities needed to escalate the dose of lenalidomide to 10 mg/day.
  Interventions: Drug: Bendamustine and Rituximab Induction followed by Rituximab and Lenalidomide Maintenance

INTERVENTIONS:
Drug: Bendamustine and Rituximab Induction followed by Rituximab and Lenalidomide Maintenance

SUMMARY:
CLL/SLL is an incurable disease with conventional chemotherapy, and there are limited treatment options available for patients who have become refractory to fludarabine- and alkylating-agent based regimens. Bendamustine is a recently FDA-approved agent with significant activity in CLL/SLL, including significant activity in the setting of fludarabine-refractory disease. However, durations of remission following bendamustine/rituximab combination therapy tend to be short in patients with heavily pre-treated disease or who have already received rituximab.

The incorporation of a maintenance therapy to overcome the shorter remission durations in this population is a reasonable and feasible option. In considering potential options for treatment of CLL/SLL as a maintenance strategy following induction chemotherapy, lenalidomide and rituximab are appealing options based on their convenient dosing schedules and recent evidence of acceptable toxicity and promising efficacy in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed CLL/SLL.
2. Understand and voluntarily sign an informed consent document.
3. Age greater than or equal to 18 years at the time of signing the informed consent document.
4. Subjects must have documented relapsed or refractory CLL/SLL.

   * Relapsed disease is defined as progressive disease after achieving a complete or partial response to the most recent therapy.
   * Refractory disease is defined as less than a partial response to the most recent therapy.
5. Subjects must have received ≥1 prior chemotherapy regimen for their disease. Prior therapy with single-agent rituximab does not meet criteria for a prior chemotherapy regimen (i.e., prior treatment must include cytotoxic chemotherapy agent).
6. In cases of SLL, subjects must have at least one bidimensionally measurable lesion at least ≥1.5 cm measured in one dimension.
7. Eastern Cooperative Oncology Group performance status of less than or equal to 2 at study entry
8. Laboratory test results within these ranges:

   * Absolute neutrophil count greater than or equal to 1500/μL
   * Platelet count great than or equal to 100,000/μL
   * Subjects with neutrophils <1500/μL or platelets <100,000/μL with splenomegaly or extensive bone marrow involvement as the etiology for their cytopenias are eligible
   * Subjects must have adequate renal function with a creatinine clearance of ≥40 mL/min as determined by the Cockcroft-Gault calculation
   * Total bilirubin less than or equal to 2X (times) upper limit laboratory normal (ULN); subjects with non-clinically significant elevations of bilirubin due to Gilbert's disease are not required to meet these criteria
   * Serum transaminases aspartate aminotransferase (AST) (SGOT) and (alanine aminotransferase) ALT (SGPT) less than or equal to 5X ULN
   * Serum alkaline phosphatase ≤5X ULN
9. Disease-free of prior malignancies for ≥2 years with the exception of basal or squamous cell skin carcinoma, carcinoma "in situ" of the breast or cervix, or localized prostate cancer (treated definitively with hormone therapy, radiotherapy, or surgery).
10. Life expectancy of at least 3 months.
11. All study participants must be willing to be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS® .
12. Subjects must not have a known history of hypersensitivity to mannitol.
13. Subjects may have received prior therapy with bendamustine or lenalidomide, but must not have disease that is refractory to bendamustine or lenalidomide.
14. Prior therapy with rituximab is permitted, even in the setting of rituximab-refractory disease.
15. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to aspirin may use warfarin or low molecular weight heparin) if clinically indicated.
16. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS® ) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

15. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.

Exclusion Criteria:

Subjects may not have received >5 lines of prior therapy for their disease. Re-treatment with an identical regimen does not count as a new regimen.

2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document or complying with the protocol treatment.

3. Pregnant or breast-feeding females. Lactating females must agree not to breast-feed while taking lenalidomide.

4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.

5. Subjects are not eligible if there is a prior history or current evidence of central nervous system or leptomeningeal involvement.

6. Use of any other experimental drug or therapy within 28 days of enrollment.

7. Known hypersensitivity to thalidomide. 8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.

9. Disease that is refractory to prior therapy with bendamustine or lenalidomide.

10. Concurrent use of other anti-cancer agents or treatments. 11. Known to be positive for HIV or infectious hepatitis (type B or C). 12. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical or breast cancer, or other cancer from which the subject has been disease free for at least 2 years.

13. Severe or life-threatening anaphylaxis or hypersensitivity reaction when previously exposed to rituximab or other monoclonal antibody therapy.

14. Chronic hepatitis B or hepatitis C infection. 15. New York Heart Association class 3-4 heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 30 months
  • The primary objective is progression-free survival for patients entering the maintenance therapy phase with rituximab and lenalidomide after induction therapy with bendamustine and rituximab. Progression is defined as radiographic or clinical progression as defined by the specified standard response criteria for Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)or initiation of a new anti-neoplastic therapy in the absence of progression. Subjects with clinical evidence of progression prior to a planned disease assessment will be evaluated at the time of clinically suspected progression.

SECONDARY OUTCOMES:
Objective Response Rates | Up to 30 months
  * Disease assessments including imaging will be performed after cycles 3 and 6 of induction chemotherapy and every 4 cycles during the maintenance portion of treatment.
  * Response and progression in cases of SLL will be evaluated using the International Working Group Criteria for response in lymphoma.38 Response and progression in cases of CLL will be evaluated in this study using the Revised International Working Group CLL 2008 Criteria for Response in CLL (IWGCLL)
  * Radiological methodologies, techniques and/or physical examination, established at baseline for the assessment and measurement of each identified lesion will be used for all subsequent assessments.
Toxicity | Up to 30 months
  • To determine toxicities observed with induction chemotherapy and maintenance therapy:
  * Safety evaluations will be based on the incidence, intensity, and type of adverse events (AEs) and clinical laboratory results.
  * Drug doses will be modified as required based on toxicity as assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Overall survival | Up to 54 months
  o Overall survival will be determined from the date of enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Chang, MD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/